CLINICAL TRIAL: NCT07238231
Title: Taiwan Preterm Infant Database: Analysis and Comparison of Birth Conditions and Exploration of Prognostic Factors
Status: Active, not recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202200008B0
Record Dates: First submitted 2025-08-29; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Preterm Infant; Full-term Infant
Keywords: Birth Conditions; Prognostic Factors
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples Without DNA — Samples Without DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- birth weight group: The cases were subdivided into three groups based on birth weight: the extremely low birth weight group (<1000 g), the very low birth weight group (1000-1500 g), and the low birth weight group (1500-2500 g).
  Interventions: Other: No Intervention: Observational Cohort
- gestational age group: The cases were subdivided into four groups based on gestational age: the extremely preterm group (<28 weeks), the early preterm group (28-32 weeks), the moderate preterm group (32-34 weeks), and the late preterm group (34-37 weeks).
  Interventions: Other: No Intervention: Observational Cohort
- combined comparison group: The cases were subdivided into twelve groups based on the cross-classification of birth weight and gestational age.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
The purpose of this study is to conduct a long-term follow-up of preterm infants with different birth conditions, aiming to provide data and resources for future care and to identify predictive and influencing factors related to their functional development over time. It is hypothesized that (1) preterm infants with varying birth conditions, such as birth weight and gestational age, will exhibit different developmental outcomes, and that the establishment of a Taiwan-specific preterm infant database is essential due to the lack of comprehensive local data and ethnic variations in gestational patterns; and (2) neonatal factors, including gestational age, birth weight, and postnatal complications (e.g., pneumonia, seizures, hypoxia), serve as potential risk factors influencing later developmental trajectories.

DETAILED DESCRIPTION:
This study uses Taiwan's Preterm Infant Database to analyze gestational age, birth conditions, and long-term developmental outcomes in preterm infants. Participants are classified by gestational age and birth weight into subgroups, with demographic, clinical, and follow-up data (e.g., Bayley-III, neurodevelopmental exams, rehabilitation records) systematically collected. All data are de-identified, coded, and validated, with confidentiality maintained under IRB oversight. Statistical methods include ANOVA, chi-square, Kruskal-Wallis, repeated-measures ANOVA, and multiple regression models to identify predictive and risk factors. Standardized procedures govern data collection, management, and analysis, with strategies to address missing or inconsistent values. This framework ensures rigor, supports predictive modeling, and provides clinically relevant insights to guide early intervention and healthcare strategies.

ELIGIBILITY:
Preterm Cases (Experimental Group)

Inclusion:

* Born <37 weeks.
* Age 0-3 years.
* Stable condition with regular outpatient follow-up, medication, and rehabilitation.

Exclusion:

* Acute illness (e.g., infection).
* Conditions affecting neurodevelopment (e.g., cerebral palsy, severe complications, pneumonia, traumatic brain injury).
* Chromosomal abnormalities.

Full-term Cases (Control Group)

Inclusion:

* Born at full term.
* Age 0-3 years.
* No disease affecting neurodevelopment.
* Caregiver consent and cooperation.

Exclusion:

* Medical diagnoses affecting neurodevelopment (e.g., traumatic brain injury).
* Neurodevelopmental disorders.
* Sensory disorders.
* Chromosomal abnormalities.

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Control and experimental group
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Bayley-III Cognitive Composite Score | Baseline
  Standardized cognitive domain score from the Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III). Scale range: higher scores indicate better cognitive development.
Bayley-III Language Composite Score | Baseline
  Standardized language domain score from the Bayley-III. Scale range: higher scores indicate better language development.
Bayley-III Motor Composite Score | Baseline
  Standardized motor domain score from the Bayley-III. Scale range: higher scores indicate better motor development.
Head Circumference | Baseline
  Head circumference measured in centimeters (cm).
Body Length | Baseline
  Body length measured in centimeters (cm).
Body Weight | Baseline
  Body weight measured in kilograms (kg).
Neurological Examination Score | Baseline
  Results from standardized neurological assessment. Scale range: higher scores indicate better neurological function.
Mobility Ability Score | Baseline
  Functional mobility assessed using age-appropriate developmental checklist. Scale range: higher scores indicate greater independence.
Presence of Medical Complications/Comorbidities | Baseline
  Recorded as a binary variable (Yes/No). Unit: Proportion (%)
Rehabilitation Participation | Baseline
  Frequency of rehabilitation sessions per week based on clinical records. Unit: Sessions per week

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD, PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan